CLINICAL TRIAL: NCT00728689
Title: A Phase I Randomized, Double-Blind, Crossover, Exploratory Study of the Pharmacokinetics of a Single Oral Dose of Form I Versus Form V Capsules of the Anti-Orthopoxvirus Compound ST-246® in Fed Normal Healthy Volunteers
Brief Title: Phase I Trial of an Investigational Small Pox Medication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SIGA Technologies (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SIGA-246-005; DMID 08-0014 (Other: NIH Contract (HHSN266200600014C))
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Results first posted 2010-02-09 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2010-09

CONDITIONS: Orthopoxviral Disease; Smallpox; Monkey Pox
Keywords: Orthopoxviral; Smallpox; Monkey pox
MeSH Terms: conditions — Smallpox; Mpox, Monkeypox | interventions — tecovirimat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group ST-246 Form I (followed by Form V) (Active Comparator): Each of six subjects receive a single oral 400 mg dose (2×200 mg) of ST-246 Form I (monohydrate) in the first intervention period, followed 10 days later (3 days post-treatment monitoring and 7 days wash-out period) in the second intervention period by a single oral 400 mg dose (2×200 mg) of ST-246 Form V (hemihydrate). Both forms of drug are orally administered within 30 minutes after a standard light meal consisting of 400-450 calories and approximately 25% fat.
  Interventions: Drug: ST-246 Days 1 - 3; Drug: ST-246 Days 11 - 13
- Group ST-246 Form V (followed by Form I) (Active Comparator): Each of six subjects receive a single oral 400 mg dose (2×200 mg) of ST-246 Form V (hemihydrate) in the first intervention period, followed 10 days later (3 days post-treatment monitoring and 7 days wash-out period) in the second intervention period by a single oral 400 mg dose (2×200 mg) of ST-246 Form I (monohydrate). Both forms of drug are orally administered within 30 minutes after a standard light meal consisting of 400-450 calories and approximately 25% fat.
  Interventions: Drug: ST-246 Days 1 - 3; Drug: ST-246 Days 11 - 13

INTERVENTIONS:
Drug: ST-246 Days 1 - 3 — First Intervention is on Days 1 - 3, and includes 6 patients dosed once orally with ST-246 Form I (Arm 1), and 6 patients dosed once orally with ST-246 Form V (Arm 2).
  Other Names: Tecovirimat
Drug: ST-246 Days 11 - 13 — Second Intervention is on Days 11 - 13 (after a 3 day post-treatment monitoring and 7 day wash-out period) where the 6 patients previously given ST-246 Form I (Arm 1) are now dosed once orally with ST-246 Form V, and the 6 patients previously given ST-246 Form V (Arm 2) are now dosed once orally with ST-246 Form I.
  Other Names: Tecovirimat

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetic parameters and safety of a single dose of ST-246 400mg Form I versus ST-246 400mg Form V capsules in fed normal healthy volunteers.

DETAILED DESCRIPTION:
This was a Phase I, double-blind, cross-over, single-dose study of the orally administered anti-orthopoxvirus compound, ST-246, to 12 healthy, fed volunteers between the ages of 18 and 50 years. Subjects were randomized such that 6 subjects received either ST-246 Form I (monohydrate) followed 10 days later after a wash-out period by Form V (hemihydrate), and 6 subjects received ST-246 Form V followed by Form I, as for the previous group.

Both forms of ST-246 were similar in the way they were manufactured. The only difference between Form I and Form V may be related to how it dissolves, and this may affect the way that it is absorbed in the human body. Information about any side-effects that may occur will also be collected in this study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 50 years
2. Available for clinical follow-up duration of study.
3. Able/willing to give written consent.
4. Good general health; no clinically significant medical history.
5. Refrain from taking any medications from screening through 72 hours after last dose.
6. Adequate venous access.
7. PE and lab results without clinically significant findings within 28 days prior to receipt of drug.
8. Meet Lab Criteria within 28 days prior to receipt of drug.
9. Negative pregnancy test
10. Non smokers
11. No alcohol or caffeine
12. Participant or partner has undergone surgical sterilization, or the participant agrees either to be abstinent or use two non-hormonal methods of contraception for duration of the study

Exclusion Criteria:

1. Marked baseline prolongation of QT/corrected QT interval (QTc) interval (
2. History of additional risk factors for Torsade de Pointes
3. Clinically significant abnormal ECG
4. Personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or prolongation of the PR interval
5. Family history of Sudden Cardiac Death not clearly due to acute myocardial infarction.
6. History of any clinically significant conditions including:

   * Asthma
   * Diabetes mellitus
   * History of thyroidectomy or thyroid disease
   * Serious angioedema episodes
   * Head trauma resulting in a diagnosis of TBI other than concussion
   * Seizure or history of seizure
   * Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with intramuscular injections or blood draws
   * Malignancy
7. Family history of idiopathic seizures
8. History or presence of neutropenia or other blood dyscrasia
9. Known Hepatitis B or Hepatitis C infection
10. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome illness.
11. Current or recent history of a clinically significant bacterial, fungal, or mycobacterial infection.
12. Known clinically significant chronic viral infection (or current clinically significant viral infection
13. History of frequent or severe headaches or migraines
14. Known chronic bacterial, mycobacterial, fungal, parasitic, or protozoal infection
15. Woman who is pregnant or is breast-feeding or planning to become pregnant
16. On any concomitant medications
17. History of drug allergy that, in the opinion of the PI, contraindicates participation in the trial.
18. Inability to swallow medication
19. Body Mass Index above 35 or below 18,
20. Current drug abuse or alcohol abuse.
21. Inability to refrain from physical exercise for a period of 24 hr before and after a PK day or refrain from consuming xanthines, grapefruit or grapefruit juice
22. Clinically significant lactose intolerance
23. Received experimental drug within 30 days
24. Vaccination within 30 days
25. Total of more than 350 milliliters (mL) of blood drawn in 2 months
26. Treatment with any immunosuppressant or immunomodulatory medication in 3 months
27. Any condition occupational reason or other responsibility that, in the judgment of the PI, would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol
28. History or diagnosis that would affect absorption of study medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Marbury, MD, Principal Investigator — Orlando Clinical Research Center
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

REFERENCES:
- [Derived] Hatmal MM, Al-Hatamleh MAI, Olaimat AN, Ahmad S, Hasan H, Ahmad Suhaimi NA, Albakri KA, Abedalbaset Alzyoud A, Kadir R, Mohamud R. Comprehensive literature review of monkeypox. Emerg Microbes Infect. 2022 Dec;11(1):2600-2631. doi: 10.1080/22221751.2022.2132882. PMID 36263798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period was approximately 2 weeks (from August 26, 2008 to September 8, 2008), plus a 30-day post-treatment follow up. The study was conducted at a Phase I Study Unit of a Clinical Research Center in Orlando, FL.
Pre-assignment Details: All participants needed to meet strict entry criteria. Sixty-three subjects were screened to randomize 12 subjects into the study.
Groups:
- ST-246 Form I Followed by Form V: Each of six subjects receive a single 400 mg dose (2×200 mg) of ST-246 Form I, followed 10 days later by a single 400 mg dose (2×200 mg) of ST-246 Form V. Both forms of drug are orally administered within 30 minutes after a standard light meal consisting of 400-450 calories and approximately 25% fat.
- ST-246 Form V Followed by Form I: Each of six subjects receive a single 400 mg dose (2×200 mg) of ST-246 Form V, followed 10 days later by a single 400 mg dose (2×200 mg) of ST-246 Form I. Both forms of drug are orally administered within 30 minutes after a standard light meal consisting of 400-450 calories and approximately 25% fat.
Period: First Intervention (Days 1 - 3)
Arm/Group | ST-246 Form I Followed by Form V | ST-246 Form V Followed by Form I
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (Days 4 - 10)
Arm/Group | ST-246 Form I Followed by Form V | ST-246 Form V Followed by Form I
Started | 6 | 6
Completed | 5 (Death in family during the Washout period. Completed First Intervention period with ST-246 Form I.) | 6
Not Completed | 1 | 0
Not completed — Death in family | 1 | 0
Period: Second Intervention (Days 11 - 13)
Arm/Group | ST-246 Form I Followed by Form V | ST-246 Form V Followed by Form I
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ST-246 Form I Followed by Form V | ST-246 Form V Followed by Form I | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (8) | 34.8 (9.4) | 34.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Secondary Outcome: Number of Study Participants Who Tolerated a Single Dose of ST-246 Form I vs. Form V as Determined by No Clinically Significant Changes in Safety Parameters
Description: Evaluated safety parameters included:
  1. physical examination/vital signs
  2. electrocardiograms (heart rate, PR interval, QRS duration, QT interval, and QTc Bazett)
  3. laboratory safety tests (hematology, chemistry, urinalysis)
  4. adverse events For a), b) and c), summary statistics (mean,SD, median, minm, maxm)for values, and changes from baseline(Day 1 pre-dose) to each timepoint, were measured and compared to laboratory normal reference ranges. Values for a)- d) were assigned grades according to DAIDS AE Grading Table. Any Grade of 3 or higher was considered severe and significant.
Time Frame: 4 weeks
Population: Both groups started with 12 particpants. Form V group lost a particpant during wash-out period due to death in the family.
Measure: Number; unit: participants
Groups:
- ST-246 Form I: ST-246 Form I administered as a single 400 mg oral dose (2×200 mg) in either first intervention period or second intervention period. Drug was administered within 30 minutes after a standard light meal consisting of 400-450 calories and approximately 25% fat.
- ST-246 Form V: ST-246 Form V administered as a single 400 mg oral dose (2×200 mg) in either first intervention period or second intervention period. Drug was administered within 30 minutes after a standard light meal consisting of 400-450 calories and approximately 25% fat.
Arm/Group | ST-246 Form I | ST-246 Form V
Number analyzed (Participants) | 12 | 11
participants | 12 | 11

2. Primary Outcome: Pharmacokinetic Parameters for a Single Dose of ST-246 Form I vs. Form V: t½
Description: Mean terminal half-life (t½; hrs) for Forms I and V were calculated from [plasma] vs time profiles.
Time Frame: Post-dose samples at 0.5,1,2,3,4,8,12,24,36,48,72 hrs
Population: Both groups started with 12 particpants. Outlier values were excluded from the half-life analyses for 3 subject PK profiles (one Form I and 2 Form V). Form V group lost a particpant during wash-out period due to death in the family.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- ST-246 Form I: ST-246 Form I administered as a single 400 mg oral dose (2×200 mg) in either first intervention period or second intervention period.
- ST-246 Form V: ST-246 Form V administered as a single 400 mg oral dose (2×200 mg) in either first intervention period or second intervention period.
Arm/Group | ST-246 Form I | ST-246 Form V
Number analyzed (Participants) | 11 | 8
hours | 27.446 (13.109) | 28.180 (21.992)
Statistical Analysis 1: Comparison: ST-246 Form I vs ST-246 Form V; A sample size of 12 subjects was chosen to provide a statistical power of 80% to detect a 25% difference of the Form V mean between the Form I and Form V doses at the 0.05 level (2-sided) for this crossover design. A parametric (normal theory) general linear model was applied and an ANOVA for a 2-way crossover design was employed to examine the differences among the 2 forms; Test type: Superiority or Other; p = 0.4591, ANOVA

3. Primary Outcome: Pharmacokinetic Parameters for a Single Dose of ST-246 Form I vs. Form V: AUC0-τ
Description: Area under the drug concentration-time curve from time zero to time t, where t is the last timepoint with a drug concentration ≥ lowest obtainable quantification (AUC0-τ; ng*hr/mL).
Time Frame: Post-dose samples at 0.5,1,2,3,4,8,12,24,36,48,72 hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ST-246 Form I | ST-246 Form V
Number analyzed (Participants) | 12 | 11
ng*hr/mL | 15624.495 (5449.188) | 20065.316 (6744.974)
Statistical Analysis 1: Comparison: ST-246 Form I vs ST-246 Form V; A sample size of 12 subjects was chosen to provide a statistical power of 80% to detect a 25% difference of the Form V mean between the Form I and Form V doses at the 0.05 level (2-sided) for this crossover design. Firstly, a parametric (normal theory) general linear model was applied and an ANOVA for a 2-way crossover design was employed to examine the differences among the 2 forms. Secondly, AUC0-τ was analyzed on a log scale, to assess bioequivalence between Form I and Form V; Test type: Superiority or Other; p = 0.0048, ANOVA

4. Primary Outcome: Pharmacokinetic Parameters for a Single Dose of ST-246 Form I vs. Form V: AUC0-∞
Description: Area under the drug concentration-time curve from time zero to infinity (AUC0-∞; ng*hr/mL).
Time Frame: Post-dose samples at 0.5,1,2,3,4,8,12,24,36,48,72 hrs
Population: Both groups started with 12 particpants. Outlier values were excluded from analyses for 3 subject PK profiles (one Form I and 2 Form V). Form V group lost a particpant during wash-out period due to death in the family.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | ST-246 Form I | ST-246 Form V
Number analyzed (Participants) | 11 | 8
ng*hr/mL | 19922.017 (6543.563) | 21982.709 (9330.953)
Statistical Analysis 1: Comparison: ST-246 Form I vs ST-246 Form V; A sample size of 12 subjects was chosen to provide a statistical power of 80% to detect a 25% difference of the Form V mean between the Form I and Form V doses at the 0.05 level (2-sided) for this crossover design. Firstly, a parametric (normal theory) general linear model was applied and an ANOVA for a 2-way crossover design was employed to examine the differences among the 2 forms. Secondly, AUC0-∞ was analyzed on a log scale, to assess bioequivalence between Form I and Form V; Test type: Superiority or Other; p = 0.0997, ANOVA

5. Primary Outcome: Pharmacokinetic Parameters for a Single Dose of ST-246 Form I vs. Form V: Cmax
Description: Maximum drug concentration in plasma, determined directly from individual concentration-time data (Cmax)
Time Frame: Post-dose samples at 0.5,1,2,3,4,8,12,24,36,48,72 hrs
Population: Both groups started with 12 particpants as 'per protocol'. Form V group lost a particpant during wash-out period due to death in the family.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ST-246 Form I | ST-246 Form V
Number analyzed (Participants) | 12 | 11
ng/mL | 1068.9 (294.3) | 1230.2 (348.6)
Statistical Analysis 1: Comparison: ST-246 Form I vs ST-246 Form V; A sample size of 12 subjects was chosen to provide a statistical power of 80% to detect a 25% difference of the Form V mean between the Form I and Form V doses at the 0.05 level (2-sided) for this crossover design. Firstly, a parametric (normal theory) general linear model was applied and an ANOVA for a 2-way crossover design was employed to examine the differences among the 2 forms. Secondly, Cmax was analyzed on a log scale, to assess bioequivalence between Form I and Form V; Test type: Superiority or Other; p = 0.0422, ANOVA

6. Primary Outcome: Pharmacokinetic Parameters for a Single Dose of ST-246 Form I vs. Form V: Tmax
Description: Time to maximum plasma concentration(Tmax; hrs) for Forms I and V were calculated from [plasma] vs time profiles.
Time Frame: Post-dose samples at 0.5,1,2,3,4,8,12,24,36,48,72 hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ST-246 Form I | ST-246 Form V
Number analyzed (Participants) | 12 | 11
hours | 3.8 (1.5) | 3.8 (1.6)
Statistical Analysis 1: Comparison: ST-246 Form I vs ST-246 Form V; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8581, ANOVA

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Twelve subjects received Form I once and 11 of the same 12 subjects received Form V once. AEs and SAEs were recorded until 72 hours and 30 days, respectively, after administration of final dose of study drug. Recording at Day 41± 2 was via phone contact. Unsolicited AEs were recorded at anytime including during the 10-day washout period.
Arm/Group | ST-246 Form I | ST-246 Form V
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 1/12 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST-246 Form I (N=12) | ST-246 Form V (N=11)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Underarm tenderness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must have sponsor's written consent to publish and must provide information to the sponsor at least 30 working days prior to publication submission deadline.